CLINICAL TRIAL: NCT05955989
Title: Relining Assessment of Digital and Conventional Fabricated Complete Denture Base
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asmaa Nabil Elboraey (Other)
Collaborators: National Research Centre, Egypt (Other)
Responsible Party: Sponsor-Investigator, Asmaa Nabil Elboraey, Associate Professor, National Research Centre, Egypt
Organization: National Research Centre, Egypt (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14860202023
Record Dates: First submitted 2023-07-10; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Problem With Dentures
Keywords: Relining; Milled denture; 3D-print; complete dentures

STUDY DESIGN:
Intervention Model Description: Three groups of completely edentulous patients. Each group will receive complete denture processed with different technique. After one year the patients will recalled and relining of the denture were made to gain the retention. After one year assessment of retention by digital force gauge, occlusion equilibrium by T-Scan and patient satisfaction (PS)
Who Masked: Participant
Masking Description: the patient is not know the type of prosthesis he will receive
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Complete denture fabricated from Conventional heat curing (Active Comparator): The patients in this group will receive complete dentures fabricated by conventional heat curing method. and they will receive soft lining of the complete dentures after one year.
  Interventions: Other: soft lining of complete denture processed by 3 different techniques.
- complete denture fabricated by CAD/CAM milled technology (Active Comparator): The patients in this group will receive complete dentures fabricated by CAD/CAM ( Computer aided design/ Computer aided manufacture) method. and they will receive soft lining of the complete dentures after one year.
  Interventions: Other: soft lining of complete denture processed by 3 different techniques.
- complete denture fabricated by CAD/CAM 3D Printed technology (Active Comparator): The patients in this group will receive complete dentures fabricated by 3D printing ( three dimension) method. and they will receive soft lining of the complete dentures after one year.
  Interventions: Other: soft lining of complete denture processed by 3 different techniques.

INTERVENTIONS:
Other: soft lining of complete denture processed by 3 different techniques. — soft lining for complete denture

SUMMARY:
The bond between the resilient denture liner material and the denture base is essential to improve complete denture accuracy and retention to the underlying ridge. The bonding characteristics between resilient denture reline materials and conventional Polymethyl methacrylate (PMMA) denture base polymers have been evaluated extensively. But with the introduction of digital fabricated complete denture, the bond characteristics between digitally fabricated dentures and denture liner is sparse.

DETAILED DESCRIPTION:
Dental prostheses fabricated using different digital technology have become popular in recent years. Computer-aided design and computer-aided manufacturing (CAD-CAM) technology provides two techniques, milled or 3D printed technique which simplified the complex dental laboratory procedures by digitalizing the prosthetic design and automating the manufacturing process. Digitally fabricated prostheses have been reported to have excellent accuracy factor that has been related to favorable clinical performance. However, bone resorption underneath any mucosa supported prosthesis is not avoidable. Resilient liners are required for most complete dentures after 6 to 12 months to improve adaptation to the underlying tissues and to reduce the force transmitted to the edentulous ridge during functionThe bond between the resilient denture liner material and the denture base is essential to improve complete denture accuracy and retention to the underlying ridge. The bonding characteristics between resilient denture reline materials and conventional Polymethyl methacrylate (PMMA) denture base polymers have been evaluated extensively. But with the introduction of digital fabricated complete denture, the bond characteristics between digitally fabricated dentures and denture liner is sparse.

Therefore, the aim of this project is to evaluate the bond strength and effectiveness of denture reline of CAD/CAM (milled and 3D printed ) fabricated complete dentures compared to conventional heat-polymerized denture base.

ELIGIBILITY:
Inclusion Criteria:

* Patients are free from any systemic diseases that might affect neuro-muscular control.
* Patients having class I maxilla-mandibular relationship
* Patients having healthy mucosa and normal salivary flow

Exclusion Criteria:

* Patients have severe bony undercut.
* Uncooperative patients.
* Patients having radiation to the head and neck region.
* Smoker patients.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of change in retentive force of the complete denture | on 3rd month of denture insertion, on 6th month of denture insertion, on the 9th month of denture insertion
  assessment of complete denture retention by digital force gauge
Assessment of change in occlusal forces during the follow up period. | on 3rd month of denture insertion, on 6th month of denture insertion, on the 9th month of denture insertion
  Assessment of occlusion equilibrium by Occlusense device

SECONDARY OUTCOMES:
Patient Satisfaction | on day one of denture insertion and on the 9th month of denture insertion ( end of the follow up period)
  a questionnaire was designed containing 5 questions regarding the following parameters: retention, comfort, appearance, phonetics and pain. Increasing the score meaning more patient satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa N. Elboraey, Asso, Prof, Principal Investigator — National Research Centre, Egypt
Locations (1):
- National Research Centre, Cairo, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No